CLINICAL TRIAL: NCT06868433
Title: Phase 1b Study of TMV Vaccine Therapy Alone and TMV Vaccine Plus Pembrolizumab for Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: TMV Vaccine Therapy Alone and With Pembrolizumab for the Treatment of Recurrent and/or Metastatic Head and Neck Squamous Cell Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Dong Shin, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006705; NCI-2024-08422 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00006705 (Other: Emory University Hospital/Winship Cancer Institute); Winship6045-23 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH); 1R01CA262123-01A1 (NIH)
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Hypopharyngeal Squamous Cell Carcinoma; Metastatic Laryngeal Squamous Cell Carcinoma; Metastatic Nasopharyngeal Squamous Cell Carcinoma; Metastatic Oral Cavity Squamous Cell Carcinoma; Metastatic Oropharyngeal Squamous Cell Carcinoma; Metastatic Sinonasal Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Nasopharyngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Recurrent Sinonasal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Unknown Primary; Stage IV Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IV Nasopharyngeal Carcinoma AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Sinonasal Cancer AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Carcinoma; Carcinoma | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; pembrolizumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (TMV vaccine therapy) (Experimental): Patients provide tissue from standard of care surgery to generate vaccine. The tumor tissue will be banked. When the patient's cancer recurs or metastasis occurs the patient will be treated as indicated. If the cancer progresses, TMV vaccine will be formulated using the banked tumor tissue. Patients receive TMV vaccine intradermally once every 2 weeks for up to 3 doses. Patients undergo echocardiography at baseline and at end of treatment and blood sample collection throughout the study. Patients may also undergo additional CT, MRI or PET on study.
  Interventions: Biological: Autologous Tumor Membrane Vesicles Vaccine; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Surgical Procedure
- Cohort 2 (TMV vaccine therapy, pembrolizumab) (Experimental): Patients provide tissue from standard of care surgery to generate vaccine. The tumor tissue will be banked. When the patient's cancer recurs or metastasis occurs the patient will be treated as indicated. If the cancer progresses, TMV vaccine will be formulated using the banked tumor tissue. Patients receive TMV vaccine intradermally once every 2 weeks for up to 3 doses. Patients also receive pembrolizumab IV on day 1 of each cycle. Cycles repeat every 3 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography at baseline and at end of treatment and blood sample collection throughout the study. Patients may also undergo additional CT, MRI or PET on study.
  Interventions: Biological: Autologous Tumor Membrane Vesicles Vaccine; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Procedure: Surgical Procedure

INTERVENTIONS:
Biological: Autologous Tumor Membrane Vesicles Vaccine — Given intradermally
  Other Names: Autologous TDMV-derived Vaccine; Autologous TMV Vaccine; Autologous TMV-based Vaccine; Autologous Tumor-derived Membrane Vesicles Vaccine
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; QL2107; RPH 075; RPH-075; RPH075; SCH 900475; SCH-900475; SCH900475
  Arms: Cohort 2 (TMV vaccine therapy, pembrolizumab)
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Surgical Procedure — Provide tissue from standard of care surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase Ib trial tests the safety, side effects and best dose of tumor membrane vesicle (TMV) vaccine therapy alone and in combination with pembrolizumab and evaluates how well it works in treating patients with head and neck squamous cell cancer that has come back after a period of improvement (recurrent) or that has spread from where it first started (primary site) to other places in the body (metastatic). Vaccines made from a person's tumor cells, such as TMV vaccines, may help the body build an effective immune response to kill tumor cells. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving TMV vaccine therapy alone or with pembrolizumab may be safe, tolerable and/or effective in treating patients with recurrent and/or metastatic head and neck squamous cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, tolerability, and recommended dose and schedule of TMV vaccine alone or TMV vaccine plus pembrolizumab in patients with surgically resected, recurrent and/or metastatic head and neck squamous cell carcinoma (HNSCC).

SECONDARY OBJECTIVE:

I. To assess vaccine-induce immune activity, antitumor response, progression-free survival (PFS) and overall survival (OS) in adult patients with recurrent and/or metastatic HNSCC administered TMV vaccine alone and TMV vaccine plus pembrolizumab.

TERTIARY/EXPLORATORY OBJECTIVES:

I. Determine whether TMV vaccine induces immune response and the magnitude of the response.

II. Next-generation sequencing (NGS) will be performed using patients' tumor samples and peripheral blood mononuclear cells to assess tumor mutational burden and identify potential neoantigens.

OUTLINE: This is a dose-escalation study of TMV vaccine alone and in combination with (fixed-dose) pembrolizumab. Patients are assigned to 1 of 2 cohorts.

COHORT 1: Patients provide tissue from standard of care surgery to generate vaccine. The tumor tissue will be banked. When the patient's cancer recurs or metastasis occurs the patient will be treated as indicated. If the cancer progresses, TMV vaccine will be formulated using the banked tumor tissue. Patients receive TMV vaccine intradermally once every 2 weeks for up to 3 doses. Patients undergo echocardiography at baseline and at end of treatment and blood sample collection throughout the study. Patients may also undergo additional computed tomography (CT), magnetic resonance imaging (MRI) or positron emission tomography (PET) on study.

COHORT 2: Patients provide tissue from standard of care surgery to generate vaccine. The tumor tissue will be banked. When the patient's cancer recurs or metastasis occurs the patient will be treated as indicated. If the cancer progresses, TMV vaccine will be formulated using the banked tumor tissue. Patients receive TMV vaccine intradermally once every 2 weeks for up to 3 doses. Patients also receive pembrolizumab intravenously (IV) on day 1 of each cycle. Cycles repeat every 3 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography at baseline and at end of treatment and blood sample collection throughout the study. Patients may also undergo additional CT, MRI or PET on study.

After completion of study treatment, patients are followed up on day 90 then every 3 weeks for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least ≥ 18 years of age
* Histologically proven squamous cell carcinoma of the head and neck (HNSCC), amenable to salvage surgery. p16 positive and negative allowed. Squamous cell carcinoma of the oral cavity, larynx, hypopharynx, oropharynx, nasopharynx, sinonasal carcinoma and cancer of unknown primary (squamous cell carcinoma only) are all allowed. They will be allowed to have up to 3 different regimens after diagnosed of recurrent or metastatic HNSCC
* Oropharyngeal tumors must have p16 or human papillomavirus (HPV) testing done
* The tumor tissues must be available and banked (- 80°C) at the time of salvage surgery (1st informed consent form [ICF] must be signed)
* Recurrent and/or metastatic HNSCC that has failed standard chemotherapy and immunotherapy. Eligible subjects must have progressed on ≥ 2 lines of standard of care prior to starting trial therapy. For patients who have relapsed within 6 months of systemic therapy given with curative intent, that therapy will count as a line of metastatic therapy. Eligible subjects will have no restriction on prior lines of therapy in the metastatic/advanced disease setting
* The tumors should be measurable by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Must have enough tissue collected after salvage surgery to make at least 3 doses of vaccine (minimum weight of the resectable tumor tissue is ≥ .5 grams) and adequate cellularity (> 40% cellularity) assessed by the head and neck pathologists
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Absolute neutrophil count ≥ 1,500 cells/uL
* Platelets ≥ 100,000/uL
* Hemoglobin ≥ 9.0g/dL (may receive packed red blood cell [prbc] transfusion)
* Total bilirubin ≤ 1.5 x the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Albumin ≥ 3.0 g/dL
* Serum creatinine ≤ 1.5 x ULN
* Calculated creatinine clearance of ≥ 50 mL/min
* International normalized ratio (INR) ≤ 1.5. Anticoagulation is allowed only with low molecular weight heparin (LMWH). Patient receiving low molecular weight (LMW) heparin on stable therapeutic dose for more than 2 weeks or with factor Xa level < 1.1U/mL are allowed on the trial
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Ability to understand and willingness to sign written informed consent documents
* Female subjects of childbearing potential must agree to use adequate contraception (e.g., hormonal or barrier method of birth control; abstinence) for the duration of study treatment and 3 months after completion
* Male subjects must agree to use adequate contraception (e.g., condoms; abstinence) for the duration of study treatment and 3 months after completion
* Female subjects of childbearing age must have a negative serum pregnancy test at study entry
* Patients who have received prior pembrolizumab are eligible

Exclusion Criteria:

* Salivary tumors and non-squamous cell histology in head and neck cancer
* Not enough tissue collected after surgery for a planned 3 doses (weight of the resectable tumor tissue is less than 1.0 gram)
* Treatment with chronic immunosuppressants (e.g., cyclosporine following transplantation)
* Prior organ allograft or allogeneic bone marrow transplantation
* Subjects with any active autoimmune disease or history of known or suspected autoimmune disease except for subjects with vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Women who are pregnant or lactating, and child-bearing potential women without adequate contraception
* Uncontrolled intercurrent illness including, but not limited to, human immunodeficiency virus (HIV)-positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study
* Clinical evidence of bleeding diathesis or coagulopathy
* Patients with prior malignancies, including pelvic cancer, are eligible if they have been disease free for > 5 years. Patients with prior in situ carcinomas are eligible provided there was complete removal
* Active bacterial or fungal infections requiring systemic treatment within 7 days of treatment
* Use of other investigational drugs (drugs not marked for any indication) within 28 days or at least 5 half-lives (whichever is longer) before study drug administration
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Non-oncology vaccines within 28 days prior to planned treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | From first dose of treatment up to 7 weeks
  DLT will be defined as treatment-related adverse event that is hematologic grade 4 or non-hematologic of grade 3 or higher severity using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. DLTs will be summarized as frequency and percentage by dose levels for cohort 1 and 2 separately.
Incidence of treatment-emergent adverse events (TEAE) | Up to 30 days after last dose of treatment
  Adverse events will be assessed and graded according to NCI CTCAE v 5.0. TEAEs will be summarized based on the number (percentage) of patients experiencing events. Summaries of treatment-related TEAEs, grade 3 or higher TEAEs, serious TEAEs, and TEAEs leading to discontinuation of study drug will be provided. TEAEs and the treatment-related TEAEs will also be summarized by severity.
Recommended phase 2 dose (RP2D) | Up to 7 weeks
  Will be determined by the principal investigator based upon all available safety and immune response data by dose levels from both cohorts 1 and 2. The RP2D may not exceed the maximum tolerated dose as estimated in cohort 2.

SECONDARY OUTCOMES:
Vaccine-induced immune response | Before and after each vaccination up to 6 weeks
  Response will be defined as the fold-change of IFNg+CD4/CD8 T cells by fluorescence activated cell sorting from peripheral blood before and after each vaccination. Summary statistics (mean, median, quartile [Q]1-Q3) will be used to describe it by dose level and time points.
Tumor response rate | Up to 12 months
  Will be assessed using Response Evaluation Criteria in Solid Tumors 1.1 criteria. Tumor response will be summarized descriptively using frequencies and percentages. Response rate will be calculated as proportion along with 95% confidence intervals using the Clopper-Pearson method.
Progression-free survival (PFS) | From start of treatment to time of progression or death up to 12 months
  PFS rates will be estimated with the Kaplan-Meier method and compared between different groups using the log-rank test.
Overall survival (OS) | From start of treatment to time of death up to 12 months
  OS rates will be estimated with the Kaplan-Meier method and compared between different groups using the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Dong M. Shin, MD, FACP, FAAAS, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Undecided